CLINICAL TRIAL: NCT03883568
Title: A 2-year Multicentre, EU, Exploratory Study Without Therapeutic Benefit in Patients With Knee Osteoarthritis to Describe, Validate, and Predict Phenotypes of Knee Osteoarthritis by Use of Clinical, Imaging, and Biochemical (Bio)Markers.
Brief Title: A 2-year, European Multicentre Study to Describe, Validate, and Predict Phenotypes of Knee Osteoarthritis
Acronym: APPROACH
Status: Completed | Type: Observational
Sponsor: F.P.J.G. Lafeber (Other)
Collaborators: GlaxoSmithKline (Industry); Nordic Bioscience A/S (Industry); University of Surrey (Other); Leiden University Medical Center (Other); Complexo Hospitalario Universitario de A Coruña (Other); Institut de Recherches Internationales Servier (Other); Newcastle University (Other); Merck KGaA, Darmstadt, Germany (Industry); Diakonhjemmet Hospital (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor-Investigator, F.P.J.G. Lafeber, Professor, director of research, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: APPROACH-OA-P01
Record Dates: First submitted 2018-07-03; First posted 2019-03-21 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: phenotypes; (bio)markers
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, blood DNA, blood RNA, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Despite a large and growing disease burden in osteoarthritis (OA), many pharmaceutical companies have abandoned OA drug development. This is mainly due to the lack of appropriate outcome measures that can robustly identify patients that can benefit from a specific therapy. Different phenotypes of OA may benefit from different types of treatment. Therefore, novel markers to identify selected phenotypes of osteoarthritis may encourage drug development.

Objective: To prospectively describe in detail pre-identified progressing phenotypes of patients with knee OA by use of conventional and novel clinical, imaging, and biochemical (bio)markers, and to validate and refine a predictive model for these (and new) progressing phenotypes based on these markers.

Study design: APPROACH is an exploratory, European, five-centre, 2-year prospective follow-up, cohort study, with extensive measurements. In this study patients are treated according to regular care by their own physician with no study related treatment prescribed. Study related diagnostic and/or monitoring procedures are applied to the patients.

Study population: Patients with tibiofemoral knee osteoarthritis, according to the clinical ACR classification criteria, pre-identified based on demographic (e.g. age), clinical (e.g. Pain NRS) and tissue structure (e.g. radiographic joint space width) parameters.

Main study parameters/endpoints: Joint tissue structure based on radiographs, MRI, and biochemical (bio)markers as well as symptoms (pain, function) and quality of life by questionnaires.

Secondary parameters: A multitude of (novel and conventional) clinical, imaging, and biochemical parameters related to osteoarthritis.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The participants will not have any direct benefit from their participation in this study other than that their OA is maximally diagnosed and followed in detail for up to 2 years (screening, baseline, 6 months, 12 months, 24 months).

DETAILED DESCRIPTION:
Patients will stay in the hospital for 4-5 hours per visit (for screening about 30 min) for physical examination, blood draw, MRI scans, radiographs of knees and hands (only at baseline and 24 months), CT scan of the knee (only at baseline and 24 months), low radiation whole body CT scan (only at baseline and 24 months), HandScan (only at baseline and 24 months), motion analysis, and performance based tests. They will be asked to fill out questionnaires about knee, hand and hip osteoarthritis, and about general health and pain. The patient council in the consortium indicated that the load is acceptable. The patient council will be involved in the execution of the study. The assumed risk is minimal for an individual patient and minimal compared to the contribution to the development of knowledge of their disease. These risks include minimal events due to blood sampling itself (such as hematoma or localized bleeding), radiation exposure by radiographic imaging techniques (with a minimal increased healthcare risk), and exposure to MRI techniques (without known risks and without use of contrast agents).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained.
2. Ambulatory (able to walk unassisted)
3. At least 18 years of age
4. Capable of understanding the study
5. Capable of writing and reading in local language
6. Predominantly tibiofemoral knee osteoarthritis and satisfy the clinical classification criteria of the American College of Rheumatology (ACR): Knee pain and three of the following criteria: over 50 years age, less than 30 minutes of morning stiffness, crepitus on active motion, bony tenderness, bony enlargement, or no palpable warmth.
7. Highest probability to progress based on the algorithm based on the following parameters:

   * Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
   * BMI (in recording height and weight)
   * Pain NRS of the index knee at the moment of the screening visit
   * Pain NRS of the index knee during the last week before the screening visit
   * Age
   * Gender
   * KIDA parameters of the index knee, based on standardized weight-bearing (KIDA) radiograph, measured < 3 months (patients with a Joint Space Width (JSW) < 2 mm of the index knee will not be included)

   Exclusion Criteria:
8. Not being able to comply to the protocol
9. Participating in a trial with local therapeutic intervention for index knee OA (pharmaceutical or surgical) or systemic Disease Modifying OsteoArthritic Drugs (DMOADs) or potential DMOADs treatments for OA at the same time or within the past 6 months or anticipated in the forthcoming; participation in non-interventional registries or epidemiological studies is allowed.
10. Surgery of the index knee in the past 6 months (to avoid interferences with imaging)
11. Scheduled or expected surgery of the index knee in the next 2 years (to avoid interferences with imaging)
12. Pregnancy (child bearing woman) because of imaging (radiation and MRI, risks)
13. Predominantly patellar femoral knee OA (clinical judgment)
14. The following secondary osteoarthritis of the knee: clinically significant deformities of the lower limbs (varus >10°, valgus >10°), septic arthritis, inflammatory joint disease, gout, major chondrocalcinosis (pseudogout), Paget's disease of the bone, ochronosis, acromegaly, haemochromatosis, Wilson's disease, rheumatic symptoms due to malignancies, primary osteochondromatosis, osteonecrosis, osteochondritis dissecans, haemophilia
15. Generalized pain syndrome, for example fibromyalgia
16. Patients with contra indication to MRI or CT
17. Hip replacement or expected hip replacement within 6 months
18. Osteosynthesis material near the knee joint
19. Self-reported severe Intervertebral disc (IVD) degeneration or facet OA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tibiofemoral knee osteoarthritis, according to the clinical ACR classification criteria, pre-identified based on demographic (e.g. age), clinical (e.g. Pain NRS) and tissue structure (e.g. radiographic joint space width) parameters.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
OA structural progression of the index knee | over two years
  radiographic joint space width in mm
OA pain progression of the index knee | over two years
  increase in points in Knee Osteoarthritis Outcome Score for pain (0-100; 0 worst, 100 best condition)

SECONDARY OUTCOMES:
OA progression of the index knee | over two years
  structural progression (e.g. cartilage volume on MRI in mm3)
OA progression | over two years
  structural progression (biochemical markers in units/ml in blood and urine)

CONTACTS AND LOCATIONS:
Overall Officials: Floris PJ Lafeber, PhD, Study Director — UMC Utrecht
Locations (5):
- Saint-Antoine hospital, AP-HP, Paris, France
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - UMC Utrecht, Utrecht
- Diakonhjemmet hospital, Oslo, Norway
- SERGAS, A Coruña, Spain

REFERENCES:
- [Derived] Jansen MP, Wirth W, Bacardit J, van Helvoort EM, Marijnissen ACA, Kloppenburg M, Blanco FJ, Haugen IK, Berenbaum F, Ladel CH, Loef M, Lafeber FPJG, Welsing PM, Mastbergen SC, Roemer FW. Machine-learning predicted and actual 2-year structural progression in the IMI-APPROACH cohort. Quant Imaging Med Surg. 2023 May 1;13(5):3298-3306. doi: 10.21037/qims-22-949. Epub 2023 Mar 10. PMID 37179936
- [Derived] Brett A, Bowes MA, Conaghan PG. Comparison of 3D quantitative osteoarthritis imaging biomarkers from paired CT and MR images: data from the IMI-APPROACH study. BMC Musculoskelet Disord. 2023 Jan 30;24(1):76. doi: 10.1186/s12891-023-06187-2. PMID 36710346
- [Derived] Roemer FW, Jansen M, Marijnissen ACA, Guermazi A, Heiss R, Maschek S, Lalande A, Blanco FJ, Berenbaum F, van de Stadt LA, Kloppenburg M, Haugen IK, Ladel CH, Bacardit J, Wisser A, Eckstein F, Lafeber FPJG, Weinans HH, Wirth W. Structural tissue damage and 24-month progression of semi-quantitative MRI biomarkers of knee osteoarthritis in the IMI-APPROACH cohort. BMC Musculoskelet Disord. 2022 Nov 17;23(1):988. doi: 10.1186/s12891-022-05926-1. PMID 36397054
- [Derived] Wirth W, Maschek S, Marijnissen ACA, Lalande A, Blanco FJ, Berenbaum F, van de Stadt LA, Kloppenburg M, Haugen IK, Ladel CH, Bacardit J, Wisser A, Eckstein F, Roemer FW, Lafeber FPJG, Weinans HH, Jansen M. Test-retest precision and longitudinal cartilage thickness loss in the IMI-APPROACH cohort. Osteoarthritis Cartilage. 2023 Feb;31(2):238-248. doi: 10.1016/j.joca.2022.10.015. Epub 2022 Nov 3. PMID 36336198
- [Derived] van Helvoort EM, Jansen MP, Marijnissen ACA, Kloppenburg M, Blanco FJ, Haugen IK, Berenbaum F, Bay-Jensen AC, Ladel C, Lalande A, Larkin J, Loughlin J, Mobasheri A, Weinans HH, Widera P, Bacardit J, Welsing PMJ, Lafeber FPJG. Predicted and actual 2-year structural and pain progression in the IMI-APPROACH knee osteoarthritis cohort. Rheumatology (Oxford). 2022 Dec 23;62(1):147-157. doi: 10.1093/rheumatology/keac292. PMID 35575381
- [Derived] Angelini F, Widera P, Mobasheri A, Blair J, Struglics A, Uebelhoer M, Henrotin Y, Marijnissen AC, Kloppenburg M, Blanco FJ, Haugen IK, Berenbaum F, Ladel C, Larkin J, Bay-Jensen AC, Bacardit J. Osteoarthritis endotype discovery via clustering of biochemical marker data. Ann Rheum Dis. 2022 May;81(5):666-675. doi: 10.1136/annrheumdis-2021-221763. Epub 2022 Mar 4. PMID 35246457
- [Derived] van Helvoort EM, Welsing PMJ, Jansen MP, Gielis WP, Loef M, Kloppenburg M, Blanco F, Haugen IK, Berenbaum F, Bay-Jensen AC, Ladel C, Lalande A, Larkin J, Loughlin J, Mobasheri A, Weinans H, Lafeber F, Eijkelkamp N, Mastbergen S. Neuropathic pain in the IMI-APPROACH knee osteoarthritis cohort: prevalence and phenotyping. RMD Open. 2021 Dec;7(3):e002025. doi: 10.1136/rmdopen-2021-002025. PMID 34911812
- [Derived] Taylor J, Dekker S, Jurg D, Skandsen J, Grossman M, Marijnissen AK, Ladel C, Mobasheri A, Larkin J, Weinans H, Kanter-Schlifke I; APPROACH research consortium and APPROACH Principal Investigators. Making the patient voice heard in a research consortium: experiences from an EU project (IMI-APPROACH). Res Involv Engagem. 2021 May 10;7(1):24. doi: 10.1186/s40900-021-00267-0. PMID 33971982
- [Derived] van Helvoort EM, van Spil WE, Jansen MP, Welsing PMJ, Kloppenburg M, Loef M, Blanco FJ, Haugen IK, Berenbaum F, Bacardit J, Ladel CH, Loughlin J, Bay-Jensen AC, Mobasheri A, Larkin J, Boere J, Weinans HH, Lalande A, Marijnissen ACA, Lafeber FPJG. Cohort profile: The Applied Public-Private Research enabling OsteoArthritis Clinical Headway (IMI-APPROACH) study: a 2-year, European, cohort study to describe, validate and predict phenotypes of osteoarthritis using clinical, imaging and biochemical markers. BMJ Open. 2020 Jul 28;10(7):e035101. doi: 10.1136/bmjopen-2019-035101. PMID 32723735